CLINICAL TRIAL: NCT05787704
Title: Walking and Thinking - Brain Activity During Complex Walking in People With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Erika Franzén, Professor, Karolinska Institutet
Other Study IDs: 4-1673/2020; 2020-03059 (Other: Ethical permit)
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Multiple Sclerosis; Gait Disorders, Neurologic; Neuro-Degenerative Disease; Aging
Keywords: functional near infrared spectrometry; gait; physical activity; cognition; brain activity
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis: People with Multiple Sclerosis, 18 years or older
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Assessment of brain activity with fNIRS and behavioural assessments (motor, motor-cognitive and cognitive) during three complex walking conditions.
  1. Dual-task walking with the auditory stroop task.
  2. Navigational walking - a course consisting of a distribution of 45 and 90 degrees turns to the left and right
  3. Navigational and dual-task walking (condition 1 and 2 together)

SUMMARY:
Every-day life means being part of a complex environment and performing complex tasks that usually involve a combination of motor and cognitive skills. However, the process of aging or the sequelae of neurological diseases such as Multiple Sclerosis (MS) compromises motor-cognitive interaction necessary for an independent lifestyle. While motor-cognitive performance has been identified as an important goal for sustained health across different clinical populations, little is known about underlying brain function leading to these difficulties and how to best target these motor-cognitive difficulties in the context of rehabilitation and exercise interventions.

The challenge of improving treatments of motor-cognitive difficulties (such as dual-tasking and navigation) is daunting, and an important step is arriving at a method that accurately portrays these impairments in an ecological valid state. The investigators aim therefore to explore brain function during complex walking in MS (in comparison with people with Parkinson's disease and healthy controls) by investigating the effects of neurological disease on motor-cognitive performance and its neural correlates during three conditions of complex walking (dual-task walking, navigation and a combination of both) using non-invasive measures of brain activity (functional near infrared spectrometry, fNIRS) and advanced gait analysis in real time in people with MS (in comparison with people with Parkinson's disease and healthy adults).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* with an MS diagnosis according to McDonald criteria
* with the ability to walk without a mobility device for ≥5 minutes continuously.

Exclusion Criteria:

* Disease or condition that affects cognition, gait or balance.
* MS relapse or change of disease-modifying treatment within the past eight weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We are studying complex walking in four different populations, people with Multiple Sclerosis, healthy young adults, healthy elderly and elderly with Parkinson's disease. We have during 2022 completed data collection (ClinicalTrials.gov ID: NCT05218213) of healthy young adults, healthy elderly and elderly with Parkinson's disease. Hence, this registration concerns the MS cohort.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Functional near infrared spectrometry (fNIRS) | During the test session during all three conditions
  The measurement of changes in concentration of HbO and HHb in the prefrontal cortex will be assessed using a NIRSPORT 2 (NIRx Medizintechnik, Berlin, Germany) device.
Gait performance during all conditions | During the test session during all three conditions
  Gait variables such as stride time and/or velocity will be analyzed with the APDM mobility system.
Dual-task performance-reaction time | During the test session during complex walking condition 1 and 3
  Cognitive performance of the dual task will be assessed as errors in the response to the Auditory stroop task.

SECONDARY OUTCOMES:
Cognitive function- composite score | During the test session, takes about 50 minutes
  The cognitive test battery comprised the following tests: The Color-Word Interference Test (CWIT), Verbal Fluency, Trail Making Test (TMT) and Ray Auditory Verbal Learning Test (RAVLT) and Symbol Digit Modalities Test (SDMT). Cognitive function will be assessed as a composite measure of these test together.
Cognitive function - verbal fluency | During the test session, takes about 12 minutes
  Verbal function, initiation & task-set switching with the Verbal Fluency test from D-KEFS (Delis-Kaplan Executive Function System).
Cognitive function - Attention and psychomotor processing speed | During the test session, takes about 3 minutes
  Attention and psychomotor processing speed will be assessed with the Trail Making Test (TMT) from D-KEFS (Delis-Kaplan Executive Function System).
Cognitive function - Episodic memory | During the test session, takes about 30 minutes
  Episodic memory will be assessed with the Ray Auditory Verbal Learning Test (RAVLT).
Cognitive function - Cognitive processing speed | During the test session, takes about 3 minutes
  Cognitive processing speed will be assessed with the Symbol Digit Modalities Test (SDMT)
Cognitive function - Inhibition & task-set switching | During the test session, takes about 5 minutes
  Inhibition & task-set switching with the The Color-Word Interference Test (CWIT) from D-KEFS (Delis-Kaplan Executive Function System).
Self-reported level of physical activity | Will be answered before the test session in the patients home or during the test session
  Assessed with the Frändin-Grimby Scale (score 1-6, higher score=better)
Physical activity level and intensity | For one week after the test session
  Assessed with accelerometers (Actigraph GT3X+)
Overall MS-disability | During the test session
  Assessed with the Expanded Disability Status Scale (EDSS). Higher scores=worse/more severe disability
Balance performance | During the test session
  Assessed with the Mini-BESTest (Balance Evaluation Systems test), 0-28p.
Anxiety and depression | Will be answered before the test session in the patients home or during the test session
  Assessed with Hospital Anxiety and Depression Scale (HADS), 0-24 on the depression and anxiety part respectively. Lower score=better
Walking ability | Will be answered before the test session in the patients home or at the test session
  Self-assessed walking ability with the WALK-12G.
Dual-task performance -errors | During the test session during dual task conditions
  Cognitive performance of the dual task will be assessed as the reaction time to respond during Auditory stroop
Disability | Will be answered before the test session in the patients home or during the test session
  WHO Disability Assessment Schedule (WHODAS) version 2.0, 12 self-assessed questions (12 to 60) more points=worse
Impact of Fatigue | Will be answered before the test session in the patients home or during the test session
  Self-assessed impact of fatigue on physical, cognitive, and psychosocial functioning, with the Modified Fatigue Impact Scale (MFIS). 21 items, scored from 0 to 4. Higher scores indicate a larger impact of fatigue.
Impact of MS on health | Will be answered before the test session in the patients home or during the test session
  Self-assessed physical and psychological impact of MS on health. 29 items, rated from 1 to 5. Higher score indicates perceived worse physical or psychological impacts of MS, respectively, on health.

CONTACTS AND LOCATIONS:
Overall Officials: Erika Franzén, PhD9, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska Institutet, Stockholm, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
The datasets generated during and/or analysed during the current study are not publicly available due to Swedish and EU personal data legislation but are available from the principal investigator on reasonable request. Any sharing of data will be regulated via a data transfer and user agreement with the recipient.
Supporting Information: SAP, Analytic Code
Time Frame: We plan to share this when applicable on OSF or similar
Access Criteria: The datasets generated during and/or analysed during the current study are not publicly available due to Swedish and EU personal data legislation but are available from the principal investigator on reasonable request. Any sharing of data will be regulated via a data transfer and user agreement with the recipient.